CLINICAL TRIAL: NCT04112836
Title: Pancreatic Cancer Malnutrition and Pancreatic Exocrine Insufficiency in the Course of Chemotherapy in Unresectable Pancreatic Cancer
Acronym: PAC-MAIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Moscow Clinical Scientific Center (Other)
Collaborators: University of Santiago de Compostela (Other); University Clinic Dr Dragisa Misovic-Dedinje (Other); University of Belgrade (Other); Hospital General Universitario de Alicante (Other); Istanbul University (Other); European Institute of Oncology (Other); IRCCS San Raffaele (Other); Bucharest Emergency Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2/2019
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Pancreatic Cancer; Exocrine Pancreatic Insufficiency; Metastatic Pancreatic Cancer; Chemotherapy; Malnutrition; Locally Advanced Malignant Neoplasm
Keywords: pancreatic cancer; locally advanced; metastatic; nutritional status; exocrine pancreatic insufficiency; chemotherapy; dose-intensity
MeSH Terms: conditions — Pancreatic Neoplasms; Exocrine Pancreatic Insufficiency; Malnutrition; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal nutritional status: Patients, fulfilled inclusion criteria with Mini-Nutritional Assessment score of 24-30 points.
- Malnourished: Patients, fulfilled inclusion criteria with Mini-Nutritional Assessment score of fewer than 17 points.

SUMMARY:
Malnutrition and cachexia are common in patients with advanced pancreatic ductal adenocarcinoma (PDAC) and have a significant influence on the tolerance and response to treatments. If timely identified, malnourished PDAC patients could be treated to increase their capacity to complete the planned treatments and therefore, possibly, improve their efficacy.

The aim of the study is to assess the impact of nutritional status, pancreatic exocrine insufficiency (PEI), and other clinical factors on patient outcomes in patients with advanced PDAC.

The nutritional status will be determined by means of Mini-Nutritional Assessment score and laboratory blood tests. PEI will be defined as the presence of typical symptoms and/or reduced fecal elastase. Analysis: chemotherapy dosing over the first 12 weeks of therapy (i.e. percent of chemotherapy received in the first 12 weeks, as defined above) PAC-MAIN will provide insights on the role of malnutrition and PEI in outcomes of PDAC.

DETAILED DESCRIPTION:
Investigators hypothesize that malnutrition has an adverse impact on the clinical course of patients with advanced PDAC treated with chemotherapy.

Aims:

To investigate the association between the nutritional status and pancreatic exocrine function and the clinical outcomes of patients with advanced PDAC.

Study design:

The PAncreatic Cancer MAlnutrition and exocrine pancreatic INsufficiency in the course of chemotherapy in unresectable pancreatic cancer (PAC-MAIN) study is a non-profit, international, multicentre, prospective, observational, cohort study evaluating the effect of the nutritional status and pancreatic exocrine function on the main outcomes of patients with advanced PDAC. The study will be carried out in Russia, Turkey, Serbia, Romania, Italy, and Spain as a part of the Pancreas 2000 Educational Program. Pancreas 2000 is a post-graduate educational program that prepares young gastroenterologists, surgeons, radiologists, and other physicians for specialization in Pancreatology.

Patient-related:

* sex, race, age at diagnosis
* Mini-Nutritional Assessment (MNA) score
* sarcopenia (measured with computed tomography (CT) fat free mass is reduced; i.e. appendicular\L2 skeletal muscle mass index <7.2 kg/m2 (men) or <5.5 kg/m2 (women));
* cachexia (weight loss (WL)>5% in last 6 months, or WL>2% if body mass index (BMI) <20 kg/m² or sarcopenia);
* 12-item functional assessment of anorexia/cachexia therapy anorexia/cachexia subscale (FAACT-A/CS-12)
* a biliary stent
* a duodenal stent
* total and direct bilirubin
* ECOG status
* European Organization for Research and Treatment of Cancer (EORTC) QLQ-PAN26 scale
* Date of diagnosis, visit 1, visit 2 (3 months), and death/loss from follow up
* Check up on survival at 6m

Tumor-related:

* Tumor site documented by endoscopic ultrasound, CT, or magnetic resonance imaging (head, body, or tail)
* Stage according to the TNM classification
* Vessels involved
* Presence and site of metastatic disease
* Ascites
* CA-19-9
* Response evaluation criteria in solid tumors (RECIST) (for visit 2)

Nutritional parameters:

* Leucocytes (lymphocytes, neutrophils), neutrophil to lymphocytes ratio, erythrocytes, hemoglobin, hematocrit, platelets
* C-reactive protein, total protein, albumin, cholesterol, iron, transferrin, ferritin, magnesium, zinc
* International normalized ratio, activated partial thromboplastin time
* Blood fasting glucose, glycated hemoglobin

Pancreatic function and treatment:

* PEI, fecal elastase-1, pancreatic enzyme replacement therapy (PERT), date of starting PERT, the dosage of daily taken PERT
* Diabetes mellitus (DM), date of DM diagnosis, DM type, DM treatment

Treatment-related:

* Planned chemotherapy protocol Dosages of chemotherapy planned (mg/m2)
* Percent of standard chemotherapy dose delivered
* Percent of planned chemotherapy delivered
* Changes to the predefined schedule (dose reduction, schedule modifications, stop before planned)
* Date of treatment start and end
* Adverse events (National Cancer Institute toxicity scale for visit 2)

Description of the intervention (schedule of visits):

Visit 1 (screening, within 1 month from initial diagnosis). Patients will be informed about the study. Once patients agree with the inclusion in the study the investigators will evaluate the inclusion and exclusion criteria. Those patients who meet all the inclusion criteria and none of the exclusion criteria will be finally included in the study. In this visit, patients, tumor-related variables, and general patients' features will be recorded, and quality of life questionnaire will be administered. The researcher will record weight, height, body mass index (BMI), unplanned WL % for the last 6 months.

Each patient's baseline nutrition status will be evaluated using the MNA scores prior to starting chemotherapy. Patients will be classified as in the group with no nutritional risk, at risk of malnutrition, or malnourished.

Nutritional parameters and pancreatic function will be evaluated through blood tests and a fecal test.

Visit 2 (3 months after the first dose of planned chemotherapy). The researcher will record in the case report form (CRF) the planned chemotherapy, schedule, doses, dose reduction, and any adverse event. The same variables recorded at Visit 1 will be checked again.

Check up 3 (end of the study, 6 months). The researcher will record in the CRF the overall survival and time until progression.

Medication of the study:

The study is of observational nature, so a pre-planned treatment is not considered. However, the use of pancreatic enzyme replacement treatment will be recorded as well as data regarding the employed chemotherapy regimen.

Power size calculation:

The expected percent of chemotherapy delivered in well-nourished patients was based on a study that assessed the chemotherapy dose intensity in gastrointestinal malignancies included pancreaticobiliary disease during the firsts 8 weeks after the start of the chemotherapy23. Based on an expected percentage of chemotherapy delivered of 70% in well-nourished patients, with a type I error of 0.05 and a type II error of 0.20, a sample size of 93 patients per group will be required in case of a percentage difference of chemotherapy delivered of 20% between well-nourished and malnourished, 163 patients per group in case of a difference of 15% between both groups and 356 patients per group in case of 10% of difference.

Discussion:

Given the sparse overall scientific data on the subject, the investigators have designed a study that addresses the impact of patient's nutritional status and dietary intervention on the clinical course of patients with advanced PDAC treated with chemotherapy and is aimed at establishing whether it affects both tolerance and tumor response to medical therapy. PAC-MAIN will be the first study specifically investigating whether the nutritional status influences the possibility to complete planned chemotherapy in patients with advanced PDAC.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* histological diagnosis of PDAC within one month from recruitment to the study;
* radiological diagnosis of the advanced stage not suitable for upfront surgical resection (either locally advanced or metastatic) within 5 weeks from recruitment to the study;
* data on the variables and the outcomes of interest are available;
* a written consent to participate in the study;
* being planned for chemotherapy;
* no past history of anticancer treatment.

Exclusion Criteria:

* poor performance status (Eastern Cooperative Oncology Group scale (ECOG) ≥ 3);
* pregnancy;
* surgery for PDAC in the past and developed progression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with unresectable locally advanced or metastatic PDAC
Sampling Method: Non-Probability Sample
Enrollment: 186 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Percent of standard chemotherapy dose delivered | 12 weeks after the diagnosis
  Drug doses will be expressed in weight-based, body surface area (BSA)-based, Area Under the Curve (AUC) units or flat dose, according to standard dosing practice for a given drug or combination. For each drug in a regimen, the sum of the doses delivered during the first 12 weeks of therapy will be divided by the sum of the expected doses based on published standard schedule and dosing. The mean percent dose delivered of all drugs in a regimen will be reported as 'percent of standard chemotherapy dose delivered.' The investigators will use percent of standard chemotherapy dose delivered to estimate the overall relative dose delivered.
Percent of planned chemotherapy delivered | 12 weeks after the diagnosis
  Similarly, the sum of the doses delivered during the first 12 weeks of therapy will be divided by the sum of the expected doses based on each patient's starting chemotherapy dose, and the mean percent dose delivered for all drugs in a regimen will be reported as 'percent of planned chemotherapy delivered.' The investigators will use percent of planned chemotherapy dose delivered to quantify further dose reductions from starting dose and as an indicator of overall toxicity.

SECONDARY OUTCOMES:
Percent of patients with chemotherapy-related toxicity in each group | 12 weeks after the diagnosis
Survival at 6 months | 12 weeks after the diagnosis, 6 months
Progression-free survival | 6 months
Quality of Life (EORTC) QLQ-PAN26 scale | 12 weeks after the diagnosis
  The pancreatic cancer module is designed for patients at all disease stages undergoing surgical resection, palliative surgical intervention, endoscopic palliation or palliative chemotherapy (Fitzsimmons et al., 1999a,b). The module comprises 26 questions assessing pain, dietary changes, jaundice, altered bowel habit, emotional problems related to pancreatic cancer, and other symptoms (cachexia, indigestion, flatulence, dry mouth, taste changes). The answers range is the following: not at all - 1 point, a little - 2 points, quite a bit - 3 points, very much - 4 points. Minimum score is 26, maximum is 106. The higher total score represents the worse quality of life.
Number of hospitalizations | 12 weeks after the diagnosis
Factors associated with the percent of chemotherapy received | 12 weeks after the diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Mariia Kiriukova, MD, Study Chair — Moscow Clinical Scientific Center
Locations (8):
- IRCCS San Raffaele Scientific Institute, Milan, Italy
- Clinical Emergency Hospital Bucharest, Bucharest, Romania
- A.S. Loginov Moscow Clinical Scientific Center, Moscow, Russia
- Serbia (2):
  - University Clinic "Dr. Dragisa Misovic-Dedinje", Belgrade
  - University of Belgrade, Belgrade
- Spain (2):
  - Alicante University General Hospital, Alicante
  - University Hospital of Santiago de Compostela, Santiago de Compostela
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kiriukova M, de la Iglesia Garcia D, Panic N, Bozhychko M, Avci B, Maisonneuve P, de-Madaria E, Capurso G, Sandru V. Pancreatic Cancer Malnutrition and Pancreatic Exocrine Insufficiency in the Course of Chemotherapy in Unresectable Pancreatic Cancer. Front Med (Lausanne). 2020 Sep 3;7:495. doi: 10.3389/fmed.2020.00495. eCollection 2020. PMID 33015088